CLINICAL TRIAL: NCT05725343
Title: A Phase III Prevention Trial of Canakinumab in Subjects at High Risk for Lung Cancer _ CANAL Study
Brief Title: A Prevention Trial of Canakinumab in Subjects at High Risk for Lung Cancer
Acronym: CANAL
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Novartis has decided to terminate the trial due to the recent results made available from the Novartis CANOPY A study (CACZ885T2301), this decision is not related to any safety data for Canakinumab
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IRFMN-LUNG-8287
Record Dates: First submitted 2022-01-12; First posted 2023-02-13 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Lung Cancer
Keywords: Lung cancer; Prevention; Canakinumab
MeSH Terms: conditions — Lung Neoplasms | interventions — canakinumab

STUDY DESIGN:
Intervention Model Description: Eligible subjects will be randomized in a 3:2 ratio to receive either canakinumab s.c. at 200 mg or placebo every two months.
Who Masked: Participant, Investigator
Masking Description: Eligible subjects will be randomized in a 3:2 ratio to receive either canakinumab s.c. at 200 mg or placebo every two months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Canakinumab (Experimental): Eligible subjects will be randomized in a 3:2 ratio to receive either canakinumab s.c. at 200 mg or placebo every two months.
  Interventions: Drug: Canakinumab
- Placebo (Placebo Comparator): Eligible subjects will be randomized in a 3:2 ratio to receive either canakinumab s.c. at 200 mg or placebo every two months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Canakinumab — Canakinumabwill be administered up to three years, or until lung cancer diagnosis, unacceptable toxicity or physician/subject's decision to withdraw, whichever comes first.
  Other Names: ilaris
  Arms: Canakinumab
Drug: Placebo — placebo will be administered up to three years, or until lung cancer diagnosis, unacceptable toxicity or physician/subject's decision to withdraw, whichever comes first.
  Arms: Placebo

SUMMARY:
Randomized phase III, double-blind, placebo-controlled, multicenter clinical trial.

DETAILED DESCRIPTION:
This is a multicentre, randomized, stratified, double-blind, placebo controlled, phase III study in subjects at high risk of lung cancer with hs CRP>3 mg/L undergoing annual screening low dose CT.

The Sponsor anticipate to screen some 6.000 subjects, of whom about 700 will be recruited and evaluated in the randomized phase 3 trial.

Eligible subjects will be randomized in a 3:2 ratio to receive either canakinumab s.c. at 200 mg or placebo every two months.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent must be obtained prior to any screening procedures.
2. Age ≥18 years and ≤75 years;
3. PLCO risk >2,5% in 6 years to undergo CT screening;
4. Annual risk of lung cancer ≥3% ( 6% at 2 years or 12% at 4 years) after the baseline CT using a second risk model which includes the presence of lung nodules such as the Brock University model;
5. CRP levels above 3 mg/L;
6. Former smokers or current smokers participating in smoking-cessation-programs or subjects with incidental diagnosis of undetermined nodules;
7. Subjects must have normal organ and bone marrow function:

   1. Haemoglobin ≥ 10.0 g/dL.
   2. Absolute neutrophil count (ANC) ≥ 1.5 x 109/L.
   3. Platelet count ≥ 100 x 109/L.
   4. Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN).
   5. Aspartate aminotransferase /Serum Glutamic Oxaloacetic Transaminase (ASAT/SGOT)) and Alanine aminotransferase /Serum Glutamic Pyruvate Transaminase (ALAT/SGPT)) ≤ 2.5 x ULN.

Exclusion Criteria:

1. Active infection;
2. Subjects with previous diagnosis of invasive cancer in the 5 years before enrolment;
3. History or evidence of tuberculosis (TB) (active or latent) infection or one of the risk factors for tuberculosis such as but not limited or exclusive to:

   1. History of any of the following: residence in a congregate setting (e.g. jail or prison, homeless shelter, or chronic care facility), substance abuse (e.g. injection or noninjection) health-care workers with unprotected exposure to subjects who are at high risk of TB or subjects with TB disease before the identification and correct airborne precautions of the subject
   2. Close contact (i.e. share the same air space in a household or other enclosed environment for a prolonged period (days or weeks, not minutes or hours)) with a person with active pulmonary TB disease within the last 12 months.
   3. Evidence of TB infection (active or latent), at Visit 1, determined by purified protein derivative (PPD) skin test and/or QuantiFERON®-TB Gold (QFT-g) assay as defined by country guidelines (refer to Determination of Tuberculosis Status, p.39).

   i. If presence of TB (active or latent) is established then treatment (according to country guidelines for TB treatment or TB treatment with immunomodulating drugs) must have been initiated or completed prior to randomization per country guidelines.

   ii. In the absence of country TB (active or latent) guidelines, the following has been demonstrated: TB has been treated adequately with antibiotics, cure can be demonstrated, and risk factors resulting in TB exposure and contracting TB have been removed (e.g. the subject does not live anymore in high TB exposure setting).
4. Subjects with suspected or proven immunocompromised state, including (a) those with evidence of Human Immunodeficiency Virus (HIV) infection; subjects on anti-retroviral therapy are excluded (b) those with any other medical condition which in the opinion of the investigator places the subject at unacceptable risk for participation in immunomodulatory therapy; or (c) those requiring systemic or local treatment with any immune modulating agent in doses with systemic effects e.g. high dose oral or intravenous steroids (> 20 mg prednisone orally daily for > 30 days, > 5 mg prednisone orally daily or equivalent dose of intravenous steroid) or high dose methotrexate (> 15 mg weekly). Topical, inhaled, local steroid use in doses that are not considered to cause systemic effects are permitted.
5. History or current diagnosis of cardiac disease, including any of the following:

   * recent myocardial infarction or coronary artery bypass graft (CABG) surgery within last 6 months,
   * uncontrolled congestive heart failure,
   * unstable angina (within last 6 months),
   * clinically significant (symptomatic) cardiac arrhythmias.
6. Known active or recurrent hepatic disorder including cirrhosis, hepatitis B and C (positive or indeterminate central laboratory results).
7. Prior treatment with canakinumab or drugs of a similar mechanism of action (IL-1β inhibitor).
8. Subjects who received any biologic drugs targeting the immune system at any time.
9. All conditions contraindicating canakinumab according to summary of product characteristics according to EMA
10. History of hypersensitivity to drugs of similar chemical classes or to canakinumab or its excipients that contraindicates the subject's participation.
11. Any life-threatening condition with life expectancy < 5 years that might prevent the subject from completing the study
12. Pregnant or nursing women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test
13. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using basic methods of contraception during dosing of study treatment and for up to 3 months after last dose of study drug. Basic contraception methods include:

    1. Total abstinence (when this is in line with the preferred and usual lifestyle of the subject). Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception
    2. Male sterilization (at least 6 months prior to screening).
    3. Barrier methods of contraception: Condom or Occlusive cap (diaphragm or cervical/vault caps).
    4. Use of oral, injected or implanted hormonal methods of contraception or other forms of hormonal contraception that have comparable efficacy (failure rate <1%), for example hormone vaginal ring or transdermal hormone contraception or placement of an intrauterine device (IUD) or intrauterine system (IUS). In case of use of oral contraception women should have been stable on the same pill for a minimum of 3 months before taking study treatment.
14. Subject with nodules larger than 8 mm with Positron emission tomography (PET) SUV >2,5 for which surgical evaluation is indicated.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2022-02-03 (Actual); Primary Completion 2022-04-03 (Actual); Study Completion 2022-09-21 (Actual)

PRIMARY OUTCOMES:
Time To Lung Cancer | date of randomization up to the date of lung cancer or, for subjects free from disease, the date of last contact, up to 48 months
  TTLC will be measured from the date of randomization up to the date of lung cancer or, for subjects free from disease, the date of last contact.

SECONDARY OUTCOMES:
Time to Lung cancer death | date of randomization, up to 48 months
  Time to Lung cancer death
Overall Survival (OS) | date of randomization, up to 48 months
  Overall Survival (OS)
cancer mortality | date of randomization, up to 48 months
  cancer mortality
shrinkage of non-solid nodules | date of randomization, up to 48 months
  shrinkage of non-solid nodules
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | date of randomization, up to 48 months
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Andrea De Censi, Principal Investigator — Ospedali Galliera di Genova
Locations (6):
- Italy (6):
  - Istituto Clinico Humanitas Rozzano, Rozzano, Milano, Italy
  - Ente Ospedaliero Ospedali Galliera, Genova
  - Ospedale San Martino, Genova
  - IRST Meldola, Meldola
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - Ospedale San Raffaele, Milan

IPD SHARING:
Plan to Share IPD: No